CLINICAL TRIAL: NCT07259668
Title: An Observational Pilot Study Evaluating the Efficacy and Safety of LPS Adsorption Using the Efferon LPS Device in Patients With Thermal Burns
Brief Title: Lipopolysaccharide Adsorption (Efferon LPS) in Patients With Thermal Burns
Status: Recruiting | Type: Observational
Sponsor: Efferon JSC (Industry)
Responsible Party: Sponsor
Other Study IDs: efferon-lps 2025-03.1
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Burns
Keywords: Hemoadsorption; Hemoperfusion; Extracorporeal therapy; LPS adsorption
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: The retrospective control group will include patients from the same medical institution's records from the previous 3 years, matched to the study cohort using propensity score matching. These patients received standard therapy for thermal burns, which could include hemofiltration or hemodiafiltration procedures.
- Baseline therapy + Efferon LPS: Patients will receive standard therapy for thermal burns treatments and Efferon LPS hemoadsorption procedure. Prospective enrollment.
  Interventions: Device: Efferon LPS

INTERVENTIONS:
Device: Efferon LPS — Efferon LPS, a medical device, which is a single-use cartridge filled with a polymeric adsorbent that selectively adsorbs endotoxin via surface-immobilized ligand and excessive cytokines via its intrinsic porosity. Two hemoadsorption procedures will be performed per patient, with a duration of 6-12 hours each and an interval of 24 hours between procedures. The procedures may be administered in combination with hemofiltration or hemodiafiltration, as determined by the investigator.
  Groups: Baseline therapy + Efferon LPS

SUMMARY:
This observational pilot study aims to establish criteria for evaluating the effectiveness of hemoadsorption with the Efferon LPS device in adult patients with burn injury. Participants will be prospectively enrolled into the treatment group and compared with a retrospectively selected control group. Each patient in the treatment group will undergo two hemoadsorption sessions, each lasting 6-12 hours, with a 24 hours interval between sessions. The procedures may be performed in combination with hemofiltration or hemodiafiltration at the investigator's discretion.

DETAILED DESCRIPTION:
Extensive burns represent a severe form of trauma that, according to the World Health Organization, cause more than 180,000 deaths worldwide each year. Despite advances in modern medicine, sepsis and other infectious complications remain leading contributors to mortality among severely burned patients.

The Efferon LPS device, originally developed for sepsis, targets both primary and secondary inflammatory mediators. This technology also shows promise in burn injury, which involves a complex systemic inflammatory response. Burn trauma induces the release of cytokines and damage-associated molecular patterns (DAMPs), while increased intestinal permeability and endotoxin translocation may lead to the appearance of pathogen-associated molecular patterns (PAMPs). Addressing both DAMPs and PAMPs is therefore essential for effective burn injury management. The aim of this study is to identify criteria for evaluating the effectiveness of hemoadsorption with the Efferon LPS device in adult patients with burn injury.

ELIGIBILITY:
Inclusion Criteria:

* Thermal burn of Ⅱ and Ⅲ severity with a lesion area of 40% or more (ICD-10: T20-T25, T29)
* Burn disease in the stage of acute toxemia or septicemia
* Frank Index ≥ 90 (Frank Index quantifies burn severity based on the depth and total surface area of the skin lesion)
* The patient's condition allows for Efferon LPS therapy for at least 6 hours

Exclusion Criteria:

* Isolated thermal inhalation injury
* Charlson Comorbidity Index > 8
* Dementia
* End-stage renal failure
* Acute pulmonary embolism confirmed by CT
* Acute myocardial infarction within the past 4 weeks
* Acute cerebrovascular accident
* Uncontrolled bleeding (acute blood loss within the past 24 hours)
* Any other condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with thermal burns undergoing treatment in State Novosibirsk Regional Clinical Hospital
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Effect of the Efferon LPS hemoadsorption on ICU length of stay | 1-28 days
  Time (days) from the start of hemoadsorption to transfer from the ICU

SECONDARY OUTCOMES:
Effect of the Efferon LPS hemoadsorption on need for vasopressor support | 1-28 days
  Need for vasopressors according to the VIS 2020 scale (Vasoactive-Inotropic Score), a weighted sum of vasoactive and inotropic medication doses; higher scores indicate greater hemodynamic support requirement (worse outcome).
Effect of the Efferon LPS hemoadsorption on pulmonary oxygen metabolic function | 1-28 days
  Value of oxygenation index (PaO₂/FiO₂ (Pa))
  Oxygenation index (PaO₂/FiO₂) = arterial oxygen partial pressure (Pa02, mmHg) / the fraction of inspired oxygen (FiO2).
Effect of the Efferon LPS hemoadsorption on duration of renal replacement therapy (RRT) | 1-28 days
  Duration of renal replacement therapy (RRT) in hours
Effect of the Efferon LPS hemoadsorption on incidence of septic complications | 1-28 days
  Frequency of septic complications
Effect of the Efferon LPS hemoadsorption on frequency of surgical interventions | 1-28 days
  Frequency of surgical interventions
Effect of the Efferon LPS hemoadsoption on 28-day mortality | 1-28 days
  Mortality rate
Effect of the Efferon LPS hemoadsoption on length of hospital stay | 1-60 days
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Igor Samatov, PhD, MD, Principal Investigator — State Novosibirsk Regional Clinical Hospital; Alexander Mezhin, PhD, MD, Principal Investigator — State Novosibirsk Regional Clinical Hospital; Vladimir Kulabukhov, PhD, MD, Principal Investigator — NV Sklifosovsky Research Institute for Emergency Medicine
Locations (1):
- State Novosibirsk Regional Clinical Hospital, Novosibirsk, Russia